CLINICAL TRIAL: NCT03336320
Title: Feasibility and Acceptability of a Web-based Multidomain Intervention With Connected Devices Made to Maintain Cognitive Function in Older Adults: a Pilot Randomised Controlled Trial
Brief Title: Feasibility and Acceptability of a Web-based Multidomain Intervention to Maintain Cognitive Function in Older Adults
Acronym: eMIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Fondation pour la Recherche Médicale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC31/17/0071
Record Dates: First submitted 2017-10-09; First posted 2017-11-08 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2021-10

CONDITIONS: Aged

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multidomain Intervention Group (Experimental): Home-based multidomain intervention composed of nutritional counselling, exercise (balance, gait, , and cognitive training provided using ICT solutions. A web platform, containing information, questionnaires, videos, games, and tests related to each one of the three components of the multidomain intervention will be made available to participants in this group.
  Interventions: Device: ICT Multidomain Intervention Training
- Control Group (Active Comparator): Participants from CG will also be equipped with wrist worn accelerometers (that will record daily activity data continuously) but contrary to MIG, participants won't have access to the password encrypted application, and therefore, to the multidomain intervention. However, they will be able to access the study website with overall information on the eMIND study and links to the website of health authorities (such as "http://www.mangerbouger.fr/PNNS" or the World Health Organization "http://www.who.int/topics/ageing/fr/") regarding healthy ageing topics. Plus, in order to control for the social aspect of MIG, participants in CG will receive monthly phone calls from the research team.
  Interventions: Device: ICT Multidomain Intervention Training

INTERVENTIONS:
Device: ICT Multidomain Intervention Training — Intervention composed of cognitive training (reasoning and memory training), nutritional counselling (advices to raise awareness about the importance of promoting a diversified and balanced diet), and physical exercises (program and monitoring of progression). The access of control group to the website will be limited to general information about eMIND study and links to the website of health authorities regarding to the healthy ageing topics.
  Other Names: Information and Communications Technologies

SUMMARY:
The primary purpose of the protocol is to evaluate the feasibility and acceptability of a home-based (using information and communication technologies) intervention composed of nutritional counselling, exercise and cognitive training in older adults and its potential effect on various health outcomes.

DETAILED DESCRIPTION:
Nutritional interventions, physical exercise and cognitive training have been used to delay cognitive decline during aging, with mixed results being obtained. However, few studies have investigated the health benefits of combining two or more of those interventions (ie, the so-called multidomain approach) in older adults. Intensive in-person multidomain intervention may difficultly be translated into the "real world" of healthcare systems because currently unpractical.

Therefore, (cost-)effective interventions provided at distance and without the physical presence of healthcare professionals have the potential to be better translatable from research to real life. Information and Communications Technologies (ICT) have a crucial role to play in this context. However, to the best of our knowledge, no studies have investigated the effects of an ICT multidomain intervention on cognition in the elderly yet.

Thus, the main objective of eMIND is to test the feasibility and acceptability of a 6-month, home-based multidomain intervention composed of nutritional counselling, exercise, and cognitive training provided using ICT solutions in people aged 65 or over.

Secondary objectives include to obtaining preliminary data on the effects of the intervention on clinical outcomes in order to inform the design and sample size calculations of a future trial.

eMIND has a mixed design, being composed of a randomized controlled trial (RCT, with two groups: the ICT multidomain intervention group vs Control Group) and a qualitative study (semi-structured interview to assess the easiness-of-use of the website).

ELIGIBILITY:
Inclusion Criteria:

* Mini-mental State Examination ≥ 24
* Presenting subjective memory complaints
* Have easy access to internet (defined as Internet access at home or elsewhere at least twice a week)

Exclusion Criteria:

* Terminal illness with life expectancy less than 6 months;
* Diagnosis of dementia of any subtype according with DSM-V
* diagnosis of neurodegenerative diseases, particularly Parkinson's disease;
* Major depression
* unstable cardiovascular condition or any other health condition that might be deteriorated by physical exercise;
* Dependency in ≥ 1 activity of daily living (basic ADL) already participating in structured sessions of physical exercise or cognitive stimulation ≥ 2 times/week in the last 2 months prior to the date of baseline assessments

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Compliance to the protocol | Assessment at the end of the intervention: 6 months after the inclusion
  Compliance to measure the feasibility of the study: Participants will be asked to connect the physical exercise interface at least twice a week, the cognitive stimulation interface at least twice a week, and the nutritional interface at least once each 15 days. Participants who adhere to >75% of this frequency of web-site use will be considered adheres (quantitative approach)
Content analysis from recorded interviews | Assessment at the end of the intervention: 6 months after the inclusion
  a content analysis from recorded interviews that will be conducted at the end of the intervention period to measure the acceptability of the trial procedures (qualitative approach)

SECONDARY OUTCOMES:
Score from MMSE | Assessment of these measures at the end of the intervention: 6 months after the inclusion
  score from MMSE
Score FCSRT | Assessment of these measures at the end of the intervention: 6 months after the inclusion
  Score from FCSRT
Score DSST | Assessment of these measures at the end of the intervention: 6 months after the inclusion
  score DSST
Score Fluency tests | Assessment of these measures at the end of the intervention: 6 months after the inclusion
  Score Fluency tests
Physical activity Monitoring | Assessment of these measures at the end of the intervention: 6 months after the inclusion
  Physical data will automatically be transferred from the wrist-worn activity monitors (Fitbit Flex 2) to the application and will generate data regarding participant's number of steps walked, energy expenditure, and walking speed, in a weekly basis
Short Physical Performance Battery | Assessment of these measures at the end of the intervention: 6 months after the inclusion
  Physical function will be evaluated by the validated short performance battery SPPB, which is based on three physical tests: timed short distance walk (4 meters at usual pace), timed repeated chair stands (5-repetition chair rise), and timed balance tests (standing balance) (20). Each of these tests is assigned a score ranging from 0 to 4, with 4 indicating the highest level of performance and 0 the inability to complete the test. A summary score ranging from 0 (worst performers) to 12 (best performers) is calculated by adding walking speed, chair stands and balance scores. From the timed short distance walk test we will calculate participants' walking speed in meters/sec; therefore, although walking speed composes the SPPB overall score, it will also be analyzed separately.
Mini-Nutritional Assessment (MNA) | Assessment of these measures at the end of the intervention: 6 months after the inclusion
  This questionnaire is composed of 18 items aiming at classifying older adults as normally nourished (24≤score≤30), at risk of malnutrition (17≤score≤23.5) or malnourished (score<17).
Health-related quality of life and Health economic Euro-QoL 5D-3L | Assessment of these measures at the end of the intervention: 6 months after the inclusion
  The health-related quality of life will be assessed by the Euro-QoL 5D-3L, a valid and short questionnaire including five questions on mobility, autonomy, daily activities, pain and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno VELLAS, Pr, Principal Investigator — Gérontopôle, CHU Toulouse
Locations (1):
- Toulouse University Hospital (CHU de Toulouse), Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andrieu S, Coley N, Lovestone S, Aisen PS, Vellas B. Prevention of sporadic Alzheimer's disease: lessons learned from clinical trials and future directions. Lancet Neurol. 2015 Sep;14(9):926-944. doi: 10.1016/S1474-4422(15)00153-2. Epub 2015 Jul 23. PMID 26213339
- [Background] Ngandu T, Lehtisalo J, Solomon A, Levalahti E, Ahtiluoto S, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H, Kivipelto M. A 2 year multidomain intervention of diet, exercise, cognitive training, and vascular risk monitoring versus control to prevent cognitive decline in at-risk elderly people (FINGER): a randomised controlled trial. Lancet. 2015 Jun 6;385(9984):2255-63. doi: 10.1016/S0140-6736(15)60461-5. Epub 2015 Mar 12. PMID 25771249
- [Background] Vellas B, Carrie I, Gillette-Guyonnet S, Touchon J, Dantoine T, Dartigues JF, Cuffi MN, Bordes S, Gasnier Y, Robert P, Bories L, Rouaud O, Desclaux F, Sudres K, Bonnefoy M, Pesce A, Dufouil C, Lehericy S, Chupin M, Mangin JF, Payoux P, Adel D, Legrand P, Catheline D, Kanony C, Zaim M, Molinier L, Costa N, Delrieu J, Voisin T, Faisant C, Lala F, Nourhashemi F, Rolland Y, Van Kan GA, Dupuy C, Cantet C, Cestac P, Belleville S, Willis S, Cesari M, Weiner MW, Soto ME, Ousset PJ, Andrieu S. MAPT STUDY: A MULTIDOMAIN APPROACH FOR PREVENTING ALZHEIMER'S DISEASE: DESIGN AND BASELINE DATA. J Prev Alzheimers Dis. 2014 Jun;1(1):13-22. PMID 26594639
- [Result] Pothier K, Soriano G, Lussier M, Naudin A, Costa N, Guyonnet S, Piau A, Ousset PJ, Nourhashemi F, Vellas B, de Souto Barreto P. A web-based multidomain lifestyle intervention with connected devices for older adults: research protocol of the eMIND pilot randomized controlled trial. Aging Clin Exp Res. 2018 Sep;30(9):1127-1135. doi: 10.1007/s40520-018-0897-x. Epub 2018 Jan 24. PMID 29368298